CLINICAL TRIAL: NCT03567538
Title: National Register Studies in Thoracic Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ulrik Sartipy, MD, PhD, MD, PhD, Karolinska University Hospital
Other Study IDs: NatRegThx
Record Dates: First submitted 2018-06-13; First posted 2018-06-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer; Pulmonary Metastasis; Surgery
Keywords: Thoracic surgery; Lung surgery; Epidemiologic Methods
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thoracic surgery — Thoracic surgery, pulmonary resection, minimally invasive thoracic surgery, video assisted thoracic surgery (VATS)

SUMMARY:
The overall project aim is to study risk and outcomes following thoracic surgery by cross-linking high-quality national Swedish health-data registers for population-based investigations of individual level clinically relevant patient data.

DETAILED DESCRIPTION:
The purpose of this research project is to study risks and outcomes in patients who underwent thoracic surgery, primarily for lung cancer. We aim to establish a fundament for the conduct of nationwide population-based studies by linking patient-level data from the Swedish quality register for thoracic surgery (ThoR) and other national health-data registers maintained by the government agencies Statistics Sweden and the National Board of Health and Welfare. Cross-linking patient-level data is possible through the Personal Identity Number assigned to every individual who has resided in Sweden on a permanent basis. The Swedish Personal Identity Number is the unique identifier in all national registers.

Specifically, we aim:

1. To analyze the association between socioeconomic factors and prognosis in patients undergoing pulmonary resection for lung cancer.
2. To investigate the implementation of minimally invasive surgery for lung cancer in Sweden.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who underwent thoracic surgery in Sweden during the study period

Exclusion Criteria:

-

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients who underwent thoracic surgery in Sweden during the study period
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 15 years
  Death from any cause

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Complications related to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Sartipy, MD, PhD, Principal Investigator — Karolinska University Hospital/Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Jackson V, Al-Ameri M, Sartipy U. Weekday and Survival After Pulmonary Resections for Lung Cancer: A Swedish Nationwide Cohort Study. Chest. 2018 May;153(5):1284-1286. doi: 10.1016/j.chest.2018.03.022. No abstract available. PMID 29731047
- [Background] Al-Ameri M, Bergman P, Franco-Cereceda A, Sartipy U. Video-assisted thoracoscopic versus open thoracotomy lobectomy: a Swedish nationwide cohort study. J Thorac Dis. 2018 Jun;10(6):3499-3506. doi: 10.21037/jtd.2018.05.177. PMID 30069346
- [Background] Al-Ameri M, Persson M, Bergman P, Franco-Cereceda A, Sartipy U. Surgery for pulmonary metastases from colorectal cancer: survival and prognostic factors. J Thorac Dis. 2018 Jun;10(6):3372-3380. doi: 10.21037/jtd.2018.05.120. PMID 30069332
- [Result] Sachs E, Jackson V, Sartipy U. Household disposable income and long-term survival after pulmonary resections for lung cancer. Thorax. 2020 Sep;75(9):764-770. doi: 10.1136/thoraxjnl-2019-214321. Epub 2020 Jun 20. PMID 32564001
- [Result] Sachs E, Sartipy U, Jackson V. Sex and Survival After Surgery for Lung Cancer: A Swedish Nationwide Cohort. Chest. 2021 May;159(5):2029-2039. doi: 10.1016/j.chest.2020.11.010. Epub 2020 Nov 17. PMID 33217414